CLINICAL TRIAL: NCT02405065
Title: Phase I Study to Assess the Safety, Tolerability and Pharmacokinetics and Anti-tumor Activity of HM95573 in Solid Tumors
Brief Title: Clinical Trial to Evaluate Safety, Tolerability and Pharmacokinetics and Anti-tumor Activity of HM95573
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-RAFI-101
Record Dates: First submitted 2015-01-15; First posted 2015-04-01 (Estimated); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HM95573 (Experimental): single arm
  Interventions: Drug: HM95573

INTERVENTIONS:
Drug: HM95573 — BID or QD, PO X 21 day cycle Number of cycles: until progression or unacceptable toxicity develops

SUMMARY:
The main objective of this study is to determine the maximum tolerated dose (MTD) and recommended phase 2 dose of HM95573.

DETAILED DESCRIPTION:
Besides the main objective, there are 3 other objectives as follows:

* To evaluate the anti-cancer effect of HM95573 in solid tumor patients
* To investigate the pharmacokinetic profile of HM95573 after oral administration.
* To investigate biomarkers related to the safety and efficacy of HM95573.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 20 years of age or older
* Subjects who have provided voluntary consent to participate in the study, and signed the written consent document.
* Estimated life expectancy of at least 12 weeks
* Histologically or cytologically confirmed advanced solid tumor

Exclusion Criteria:

* Symptomatic or uncontrolled central nervous system metastases
* Patients who are unable to take tablets orally or have a clinically significant gastrointestinal disorder, which may interfere with administration, metabolism and absorption of the investigational drug.
* Patients who, in the investigator's opinion, are not suitable for the study for any other reason.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-01-12 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2018-05-16 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Dose limiting Toxicity will be evaluated on Day 28 during Cycle 1

SECONDARY OUTCOMES:
Overall rsponse rate | 6-12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yohan Kim, MD, Study Director — Hanmi Pharmaceutical co., ltd.
Locations (1):
- Hanmi Clinical, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided